CLINICAL TRIAL: NCT02616900
Title: eQUEST -- ESIGHT QUALITY OF LIFE AND EFFICACY STUDY A Multi-center, Prospective Cohort Study to Assess the Impact of eSight Eyewear on Functional Vision Improvement and Quality of Life in a Low Vision Population
Brief Title: eSight Eyewear Quality of Life and Efficacy Study
Acronym: eQUEST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: eSight Corporation (Industry)
Collaborators: Johns Hopkins University (Other); Université de Montréal (Other); University Health Network, Toronto (Other); Vitreous and Retina Consultants PA (Unknown); University of Michigan (Other); Bascom Palmer Eye Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 00014027
Record Dates: First submitted 2015-11-23; First posted 2015-11-30 (Estimated); Results first posted 2019-04-05 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Vision, Low
MeSH Terms: conditions — Vision, Low

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- eSight Eyewear (Experimental): Main arm
  Interventions: Device: eSight Eyewear

INTERVENTIONS:
Device: eSight Eyewear — primary intervention

SUMMARY:
The "eSight Quality of Life and Efficacy Study" (eQUEST) is a prospective cohort study intended to demonstrate the functional vision and Quality of Life (QoL) improvement provided by eSight Eyewear to persons with significant visual impairment resulting from various eye conditions. The multi-site study will evaluate the efficacy of the eSight device for various Activities of Daily Living (ADLs) across a broad range of subject ages and disease types.

DETAILED DESCRIPTION:
Subjects will receive an initial benchmark assessment to determine their visual function. This includes standard clinical tests for acuity and contrast performance. Subjects will then receive a demonstration of the device. If the demonstration shows favourable results (improved functional visual performance for some rudimentary tasks such as reading), and the subject consents to the study, the subject will return to the site a week later to receive their personalized device (lens prescriptions incorporated into the unit), and more comprehensive training on its operation. They will then use the unit in their home/work/school environment over a period of three months. At the start of the study, after a period of one month, and at the end of the three month period, the subject will visit the clinical setting for administration of various specified ADL tasks, and the Veterans Affairs (VA) Low Vision (LV) Visual Function Questionnaire (VFQ) 48-question VA LV VFQ-48 survey. The intent of this repetition is to understand how ADL proficiency and VFQ-48 QoL assessment changes over time, as the subject becomes more accustomed to the device.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects between the ages of 13-75.
2. Subjects have been diagnosed with one of the following low vision conditions: Diabetic Retinopathy, Stargardt's Disease, Age Related Macular Degeneration, Leber's Disease, Retinopathy of Prematurity, Cone Rod Dystrophy, or Ocular Albinism .
3. Subject must have distance Best Corrected Visual Acuity (BCVA) measured with Early Treatment Diabetic Retinopathy Study (ETDRS) chart of between 20:60 and 20:400 in the better eye.
4. Subject must have a functional field of view of at least 20 degrees (bilateral or monocular). Field need not be centrally located.
5. If the subject is employed, they must be prepared to use eSight Eyewear in their workplace environment, have informed their employer of their involvement in the study, and received permission from their employer to bring eSight Eyewear into the workplace. If the subject is self-employed, they must be prepared to use eSight Eyewear in their workplace environment. Similarly if the subject is a student, they must be prepared to use eSight Eyewear in their educational environment.
6. Subject must be, in the opinion of the examiner, highly motivated, alert, articulate, mentally competent and able to understand and comply with the requirements of the study (defined herein).
7. Subject must provide informed consent. Subjects under the age of majority must have a legal guardian present during the informed consent process, who must sign the Informed Consent form on their behalf.
8. Subject must agree to use eSight Eyewear only under conditions that will not jeopardize the safety of either the user or the device.

Exclusion Criteria:

1. Subject must not be currently undergoing any medical or surgical procedures resulting in unstable vision.
2. Subjects for whom their vision, for whatever reason, can be considered unstable.
3. Subjects who have undergone cataract, refractive, or other surgical procedures related to vision in the six month period prior to the study.
4. Subjects who have undergone any eyesight-related injections (e.g. anti-VEGF) in the two month period prior to the study because of active bleeds in the retina. Ongoing anti-VEGF treatments are permitted if subject is in a "Treat and Extend" or pro re nata ("PRN") disease management, and macula is dry.
5. Subjects unable or unwilling to adhere to the examination schedules as they are described in the study protocol. This may also include Subjects already enrolled who, for whatever reason become unable or unwilling to continue the study. This may also include subjects for whom the travel time to/from the study site is unacceptable.
6. Subjects who self report a history of alcoholism, drug abuse or psychosis, Subjects who exhibit clinical evidence of depression, poor motivation, emotional or intellectual problems, or any other conditions which would likely limit validity of consent or appropriate responses to participate in the study or who are deemed unsuitable psychologically or physiologically for study participation by the investigator.
7. Subjects who may have a conflict of interest with eSight Corp, which could reasonably influence their participation in the study.

Ages: 13 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2015-12-16 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (4):
  - Vitreous and Retina Consultants PA, Lakeland, Florida
  - Lighthouse For the Blind of the Palm Beaches, West Palm Beach, Florida
  - Johns Hopkins University School of Medicine, Wilmer Eye Institute, Baltimore, Maryland
  - University of Michigan Kellogg Eye Center, Ann Arbor, Michigan
- Canada (2):
  - Toronto Western Hospital, Toronto, Ontario
  - Université de Montréal, School of Optometry, Montreal, Quebec

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 51 participants selected from the patient population at six low vision rehabilitation clinics, in the period Dec 16, 2015 through September 19, 2016.
Pre-assignment Details: The study had only one arm.
Period: Overall Study
Arm/Group | eSight Eyewear
Started | 74
Completed 3mo Trial | 57
Completed | 51 (Six participants not included in study results because of incomplete data.)
Not Completed | 23
Not completed — Lack of Efficacy | 7
Not completed — Lost to Follow-up | 2
Not completed — Protocol Violation | 5
Not completed — Withdrawal by Subject | 3
Not completed — Incomplete data | 6

BASELINE CHARACTERISTICS:
Arm/Group | eSight Eyewear
Number analyzed (Participants) | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3
  Between 18 and 65 years | 39
  >=65 years | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (17.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Quality of Life Improvement After Three Months of Device Use
Description: The study seeks to quantify, after a period of usage of the device of three months, improvement in subjects' Quality of Life using the validated tool, "Veterans Affairs (VA) Low Vision (LV) Visual Functioning Questionnaire (VFQ) - 48 Questions" (VA LV VFQ-48). Quality of Life is measured in Logits. Individual scores ranged from -5 to +10 (a higher number is a better score). Overall improvement was 0.84 Logits.
Time Frame: Baseline and after three months of device use.
Measure: Mean (Standard Deviation); unit: Logits
Arm/Group | eSight Eyewear
Number analyzed (Participants) | 51
Logits | 0.84 (1.265)

2. Secondary Outcome: Improvement in Visual Acuity
Description: The study seeks to quantify, after a period of usage of the device of three months, improvement in visual acuity using standard optometric charts (e.g. "20/400 to 20/160", etc.). We measured LogMAR acuity on a standard ETDRS chart. Results show an average greater than seven-line improvement (-0.76 LogMAR).
Time Frame: Baseline and after three months of device use.
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | eSight Eyewear
Number analyzed (Participants) | 51
LogMAR | -0.76 (0.30)

3. Secondary Outcome: Improvement in Visual Contrast Performance in Log Units.
Description: The study seeks to quantify, after a period of usage of the device of three months, improvement in contrast performance using a standard optometric "Mars Contrast Chart". Outcome is measured in Log Units ranging from 0.04 to 1.92 in decrements of 0.04 log units, a higher score indicating better contrast performance. The scale of the Mars Contrast Chart is interpreted as follows:
  0.0 - 0.5 Log Units: Profound Loss 0.5 - 1.0 Log Units: Severe Loss 1.0 - 1.5 Log Units: Moderate Loss 1.5 - 1.75 Log Units: Normal Vision (>60yrs) >1.75 Log Units: Normal Vision (<60yrs)
Time Frame: Baseline and after three months of device use.
Measure: Mean (Standard Deviation); unit: Log Units
Arm/Group | eSight Eyewear
Number analyzed (Participants) | 51
Log Units | 0.53 (0.55)

ADVERSE EVENTS:
Time Frame: 54 weeks. January 20, 2016 - February 6, 2017
Description: All-Cause Mortality, Serious, or Other (non-serious) Adverse Events were monitored/assessed, but none observed. We define an adverse event as any event whereby patient health or safety is adversely affected in any manner by the study device.
Arm/Group | eSight Eyewear
All-Cause Mortality (participants affected / at risk) | 0/74
Serious Adverse Events (participants affected / at risk) | 0/74
Other Adverse Events (participants affected / at risk) | 0/74

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-21): https://cdn.clinicaltrials.gov/large-docs/00/NCT02616900/Prot_SAP_000.pdf